CLINICAL TRIAL: NCT02163863
Title: BioMimics 3D Stent Clinical Investigation: The Mimics Study
Acronym: Mimics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veryan Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mimics
Record Dates: First submitted 2014-06-09; First posted 2014-06-16 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral arterial disease (PAD); Peripheral vascular disease (PVD); Biomimetic stent; Helical centerline
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BioMimics 3D (Experimental): The BioMimics 3D Stent System, delivering a self-expanding Nitinol stent with 3D helical centerline geometry.
  Interventions: Device: Femoropopliteal stenting
- Control (Active Comparator): CR Bard LifeStent System, delivering a self-expanding Nitinol stent
  Interventions: Device: Femoropopliteal stenting

INTERVENTIONS:
Device: Femoropopliteal stenting

SUMMARY:
Primary purpose of the Mimics Study is to evaluate the safety and performance of the BioMimics 3D Stent System in the treatment of symptomatic SFA/proximal popliteal disease.

DETAILED DESCRIPTION:
The Mimics Study is a prospective, part randomized study; an initial roll-in registry of 10 subjects treated with BioMimics 3D followed by a randomized assignment to treatment with BioMimics 3D or Control on a 2:1 basis for 76 subjects.

The primary purpose of the study is to evaluate the safety and performance of the BioMimics 3D Stent System in the treatment of symptomatic SFA/proximal popliteal disease based on:

* Safety; measured by freedom from major adverse events determined at 30 days after the procedure, compared to historic controls.
* Performance; measured by freedom from clinically driven TLR at 6 months, compared to historic controls.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* The subject or legal guardian has been informed of the nature of the study and agrees to its provisions and has provided informed written consent
* The subject is willing to be available for the appropriate follow-up for the duration of the study
* Rutherford 1-4(mild claudication to ischemic rest pain), with an occlusion or de novo and/or restenotic SFA/PPA lesion ≥50% and ABI/TBI <0.90/0.80
* Single target lesion located at least 1 cm distal to the take-off of the profunda femoris artery and at least 3 cm proximal to the highest point of the cortical margin of the femur
* Target vessel reference diameter is ≥3.5 mm and ≤7.0 mm
* Target lesion length is ≥4.0 cm and ≤10.0 cm, and must be intended to be covered with one single stent only. A second stent is permitted to be placed only if, in the physician's opinion, the first stent did not achieve an optimum clinical result
* Adequate distal run-off to the ankle in the target limb (defined as having at least one patent calf vessel <50% stenosed
* Life expectancy >24 months

Exclusion Criteria:

* Women who do not have a negative serum or urine pregnancy test documented within 7 days prior to enrollment (if not already post menopausal) or women who do not agree to use an adequate birth control method for up to 24 months after Device implantation
* An uncontrolled infectious disease
* A condition that inhibits radiographic visualisation of the arteries
* Any condition that precludes safe access with PTA devices, such as: excessive common femoral artery disease, unresolved fresh thrombus in the target lesion/vessel, or a target lesion/vessel that is excessively tortuous or calcified
* Known allergy to, or intolerance of, Nitinol
* Known intolerance of aspirin and/or clopidogrel
* Known hypersensitivity to contrast media which cannot be pre-treated
* Participation in another device or drug study. Subject must have completed the follow- up phase of any previous study at least 30 days prior to enrollment into this study. The subject may only be enrolled in this study once
* The subject is unable and/or unwilling to cooperate with study procedures or required follow-up visits
* History of bleeding diatheses or coagulopathy or will refuse blood transfusions
* Known impaired renal function, defined as creatinine >2.5 mg/dl except subjects under chronic renal replacement therapy
* Known platelet count <80,000 cells/mm3 or >700,000 cells/mm3
* Known WBC of <3,000 cells/mm3
* The subject is unable to bend lower limbs (full knee flexion) and/or has a knee prosthesis
* Previous treatment of the target lesion 6 months prior to enrollment; previous femoropopliteal bypass in the target vessel; previous stenting of the target lesion
* Previous stenting of the SFA, popliteal and tibial arteries within the target limb
* Target lesion located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion
* Target lesion requires treatment other than standard PTA prior to stent placement (i.e., no other devices or procedures such as cutting balloons and laser atherectomy are permitted to be used during the index procedure)
* Lesions in contralateral SFA that require intervention during the index procedure, or within 30 days after the index procedure, unless both limbs are able to be and are included in the study
* Multiple lesions in the target vessel that require stenting within 30 days after study procedure
* Target lesion length is > 10cm or the physician believes prior to stent placement that the lesion cannot be covered by one single stent
* The target lesion is severely calcified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-02; Primary Completion 2012-10 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Primary safety endpoint | 30 days
  Freedom from major adverse events defined as death, amputation and target lesion revascularization (TLR)
Primary performance endpoint | 6 months
  Freedom from clinically driven TLR

SECONDARY OUTCOMES:
Acute procedural outcomes | Within 30 days of the procedure
  * Device deployment success
  * Acute procedural success
  * Procedural complications
Post implant anatomical outcomes | Immediately post implant but within the index procedure
  - Stented vessel geometry, i.e. presence/absence of 3D helical geometry in the stented region
Mechanical outcomes | 30 days, 6, 12 and 24 months
  - Stent integrity, i.e. presence/absence of kinks and fractures
Haemodynamic outcomes | discharge, 30 days, 6, 12 and 24 months
  * Restenosis measured by duplex ultrasound and angiography.
  * Swirling flow
Clinical and functional outcomes | discharge, 30 days, 6, 12 and 24 months
  * Rutherford classification (not at discharge)
  * ABI
  * Walking impairment questionnaire (not at discharge)
  * Freedom from major adverse events at 30 days, 6, 12 and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, M.D., Principal Investigator — Universitäts-Herzzentrum Freiburg Bad Krozingen; Sebastian Sixt, MD, Principal Investigator — Medizinisches Versorgungszentrum Hamburg; Henrik Schroeder, MD, Principal Investigator — Zentrum für Minimal Invasive Therapie Berlin; Horst Sievert, MD, Principal Investigator — Cardiovascular Center Frankfurt; Karl-Ludwig Schulte, MD, Principal Investigator — Königin Elisabeth Herzberge Berlin; Gunnar Tepe, MD, Principal Investigator — Klinikum Rosenheim; Giovanni Torsello, MD, Principal Investigator — St. Franziskus Hospital Münster; Dierk Scheinert, MD, Principal Investigator — Park-Krankenhaus Leipzig
Locations (1):
- Universitaets-Herzzentrum Freiburg-Bad Krozingen, Bad Krozingen, Germany

REFERENCES:
- [Result] Zeller T, Gaines PA, Ansel GM, Caro CG. Helical Centerline Stent Improves Patency: Two-Year Results From the Randomized Mimics Trial. Circ Cardiovasc Interv. 2016 Jun;9(6):e002930. doi: 10.1161/CIRCINTERVENTIONS.115.002930. PMID 27208046